CLINICAL TRIAL: NCT06491771
Title: A Randomized Split-face Study of a Precision Cryotherapy Via Boosting Mode Combined With Tranexamic Acid Versus Normal Saline in the Treatment of Melasma
Brief Title: A Cryotherapy With Tranexamic Acid Versus Normal Saline in the Treatment of Melasma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Prof. Dr., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si 477/2024
Record Dates: First submitted 2024-06-25; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Cryotherapy Effect

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- cryotherapy with tranexamic acid (Active Comparator): precision cryotherapy via boosting mode combined with tranexamic acid
  Interventions: Device: TargetCool
- cryotherapy with normal saline (Placebo Comparator): precision cryotherapy via boosting mode combined with normal saline
  Interventions: Device: TargetCool

INTERVENTIONS:
Device: TargetCool — The patients were treated with TargetCool via boosting mode combined with tranexamic acid and normal saline on each side of cheek for 4 times every 1 week

SUMMARY:
This study aimed to evaluate the effectiveness of a precision cryotherapy via boosting mode combined with tranexamic acid versus normal saline in the treatment of melasma. Eighteen patients aged 25 to 60 years diagnosed with epidermal-typed melasma sized equal to or more than 2 cm on both cheeks were included. The patients were treated with a precision cryotherapy via boosting mode combined with tranexamic acid and normal saline on each side of cheek for 4 times every 1 week. Then, they were follow up at 1 and 3 months after the last treatment. Subjective assessment of physician and patient improvement were evaluated. Moreover, Melasma Area and Severity Index (MASI), melanin and erythema index using Mexameter were also recorded.

DETAILED DESCRIPTION:
TargetCool via boosting mode combined with tranexamic acid versus normal saline were studied in patients diagnosed with epidermal-typed melasma.

ELIGIBILITY:
Inclusion Criteria:

* The patients diagnosed with epidermal-type melasma sized equal to or more than 2 cm on both sides of cheeks
* Fitzpatrick skin type II-IV

Exclusion Criteria:

* Pregnant or lactation
* Subjects who have been treated with any kind of energy-based device 6 months prior to the inclusion
* Subjects who have been treated with topical or oral treatment for melasma 6 months prior to the inclusion
* Subjects who allergy to cryotherapy such as cryoglobulinemia, cold urticaria, and abnormal cold tolerance
* Subjects with abnormal sensation such as diabetes mellitus
* Active skin infections
* History of hypertrophic scars or keloids History of hypertrophic scars or keloids

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The change of Melasma Area and Severity Index score | Baseline, 1, 2, 3 weeks after the first treatment and 1, 3 months after the last treatment
  Two blind dermatologists evaluated Melasma Area and Severity Index score on each side of cheek in every visits (0-48; best to worse)

SECONDARY OUTCOMES:
Physician improvement score | 1, 2, 3 weeks after the first treatment and 1, 3 months after the last treatment
  Using quartile scale (<0% = worsen; 0% = no change; 1-25% = mild improvement; 26-50% = moderate improvement; 51-75% = marked improvement; 76-100% = complete improvement)
Overall improvement by patients | 1, 2, 3 weeks after the first treatment and 1, 3 months after the last treatment
  Using quartile scale (<0% = worsen; 0% = no change; 1-25% = mild improvement; 26-50% = moderate improvement; 51-75% = marked improvement; 76-100% = complete improvement)
the changes in melanin index | Baseline, 1, 2, 3 weeks after the first treatment and 1, 3 months after the last treatment
  Using Mexameter
the changes in erythema index | Baseline, 1, 2, 3 weeks after the first treatment and 1, 3 months after the last treatment
  Using Mexameter
Side effects | Baseline, 1, 2, 3 weeks after the first treatment and 1, 3 months after the last treatment
  After treatment on both sides

CONTACTS AND LOCATIONS:
Overall Officials: Woraphong Manuskiatti, MD, Principal Investigator — Mahidol University
Locations (1):
- Department of Dermatology, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No